CLINICAL TRIAL: NCT04120324
Title: Incidence of 30 Day Return to Hospital Following Same Day Discharge Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Donald J Young, MD, FRCPC, Clinical Associate, University of British Columbia
Other Study IDs: H19-02526
Record Dates: First submitted 2019-09-29; First posted 2019-10-09 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis, Hip; Arthroplasty Complications; Complication of Surgical Procedure; Perioperative Complication
Keywords: complication; surgery
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Eligibility Determination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Eligible & Discharged Same Day: Surgeon earmarks patient as potentially eligible for Same Day Discharge. Preoperative Assessment by Physiotherapy and Anesthesia confirms patient is Same Day Discharge eligible. Patient undergoes Primary Single Joint Total Hip Arthroplasty and is discharged home on the day of surgery.
  Interventions: Other: Eligible for Same Day Discharge; Procedure: Primary Single Joint Total Hip Arthroplasty; Other: Discharge Same Day
- Eligible but NOT Discharged Same Day: Surgeon earmarks patient as potentially eligible for Same Day Discharge. Preoperative Assessment by Physiotherapy and Anesthesia confirms patient is Same Day Discharge eligible. Patient undergoes Primary Single Joint Total Hip Arthroplasty but is NOT discharged home on the same day as the surgery, and remains in hospital for a minimum of one night following surgery. Reasons for not being discharged same day include potential problems related to Surgery (eg. complication), Anesthesia (eg. prolonged effect), or patient factors (egs. pain, nausea, mobility difficulties, etc.).
  Interventions: Other: Eligible for Same Day Discharge; Procedure: Primary Single Joint Total Hip Arthroplasty
- Not Eligible for Discharge Same Day: Surgeon earmarks patient as potentially eligible for Same Day Discharge. Preoperative Assessment by Physiotherapy and/or Anesthesia deems the patient to NOT be eligible for Same Day Discharge. The patient undergoes Primary Single Joint Total Hip Arthroplasty and remains for a minimum of one overnight in hospital following hip replacement surgery.
  Interventions: Procedure: Primary Single Joint Total Hip Arthroplasty

INTERVENTIONS:
Other: Eligible for Same Day Discharge — Preoperative Physiotherapy and Anesthesia Criteria met.
  Groups: Eligible & Discharged Same Day; Eligible but NOT Discharged Same Day
Procedure: Primary Single Joint Total Hip Arthroplasty — Total Hip Replacement Surgery
Other: Discharge Same Day — Postoperative criteria for Same Day Discharge met.
  Groups: Eligible & Discharged Same Day

SUMMARY:
Amongst patients who are discharged home from hospital on the same day as their elective Primary Total Hip Arthroplasty, the Investigators seek to quantify the incidence of return to hospital within 30 days of surgery for assessment &/or treatment of surgical related problems or complications. This incidence rate will be compared to a cohort of patients who are not discharged on the same day as their Primary Total Hip Arthroplasty. The Investigators wish to know if the incidence of 30 day return to hospital is significantly different between these two groups of patients.

DETAILED DESCRIPTION:
At UBC Hospital, a program to facilitate same day discharge of elective Primary Total Hip Arthroplasty patients was developed in 2017/18. The program is called the "Short Term Accelerated Recovery" (STAR) program, and patients within the program are called "STAR Patients." The first patient in the program had their surgery on Oct 15, 2018, and the program has been running ever since.

The STAR process begins by the attending surgeon (there are 5 Arthroplasty Surgeons at UBC involved in this program) earmarking a patient as a potential same day discharge candidate based on their assessment of the patient. Following this, the patient is assessed by both Physiotherapy and Anesthesia to either confirm or reject their STAR eligibility.

STAR eligibility criteria can be divided into both Social and Clinical requirements. The Social requirements are for the patient to live within an hour's drive of the Vancouver General Hospital (VGH) Emergency Room, and that they have a support person (either family or friend) that will stay with them in their home for at least the first 24 hours following surgery and can be called upon at any time subsequent to help in caring for the patient or facilitating their return to hospital if needed.

Strict Clinical Requirements to be STAR Eligible were established by the Dept of Anesthesia based on best evidence and expert opinion. These criteria were used to establish a "Check-List" of items to ensure all eligibility criteria are met. Items on this Checklist included the correct Surgical Procedure, patient age ≤ 75, Pre-Anestheic Risk Assessment, and Lab Result Reviews.

Patients initially enrolled in the STAR Program by their Orthopedic Surgeon at the time of surgical booking [presently a total of 87 patients] could end up in one of three possible cohorts following their surgery:

1. The patient was deemed STAR eligible preoperatively, had their hip replacement surgery and went home the same day as their surgery [presently 24 patients].
2. The patient was deemed STAR eligible preoperatively, had their hip replacement surgery but were NOT sent home same day as their surgery for failing to meet criteria for safe discharge and thus staying a minimum of one overnight in hospital [presently 24 patients].
3. The patient was deemed NOT eligible for STAR prior to their surgery, and therefore stayed at least one night in hospital following their surgery [presently 39 patients].

Thus far, the STAR program has failed to adequately assess the incidence of 30 day post-surgical complications. Despite an infrastructure to attain this quality assessment being in place by way of a postoperative survey sent to patients via Email, return of these surveys has been minimal thus far. As a result, the Investigators are seeking a more robust and comprehensive search of postoperative hospital encounters for surgically related problems amongst these patients by way of chart review.

This project is a retrospective cohort quality assurance chart review study. Given that the criteria for enrollment in STAR is site specific and has not been established before, this project is designed to be both a preliminary safety assessment and also able to inform future prospective studies on the program's safety for potential sample sizes needed for such assessments. As well, the study would also expose the potential for a higher than expected return to hospital for same day discharge patients which may not otherwise have been known.

A log of all patients initially enrolled as potentially "STAR Eligible" by their surgeon has been maintained by the PI. Using this list of patients, the following sequence of events will occur to assess each for hospital encounters for surgical related problems, inquiries or complications during the 30 days immediately following surgery:

1. All patient's charts, both paper records at VGH and UBC Hospital, as well as electronic charts within the BC Care Connect network that can show encounters at hospitals throughout the province of British Columbia, will be retained by Research Personnel.
2. Charts will be perused for any hospital encounters during the 30 days immediately post the date of surgery.
3. If encounters are found, the specific nature of the encounter will be ascertained.
4. Study personnel will decide, based on the clinical presentation and documentation available on the patient's chart, whether the encounter may be considered a "surgically related problem, inquiry or complication".

   Examples of surgically related problems include (but are not limited to) wound or surgical site infection, deep vein thrombosis, pneumonia, urinary tract infection, pain issues as a result of having surgery, failure or concerns for the function of the new prosthesis, trauma or falls as a result of reduced mobility following surgery.
5. Some encounters may be obvious as surgically related problems - eg. concerns for a possible wound infection at the surgical site. Others may be less obviously surgically related depending on the presentation - eg. sepsis or organ failure. It will be left to the PI to invigilate and decide whether the reasons for hospital encounter are or are not obviously surgical in nature. For those deemed not obviously surgical, opinion will be sought from 2 independent specialists in Perioperative Internal Medicine on whether they feel the encounters to be related to the patient's hip arthroplasty. Reviewers will be blinded to each other's opinions. If both Reviewers agree that the encounter was for a surgically related problem then it will be tallied as such. If there is disagreement or both believe the problem to not be surgically related then it will not be considered a surgically related hospital encounter.
6. If a hospital encounter is found amongst the patient's records, but no documentation about the nature of the encounter is available, then the Patient's Orthopedic Surgeon will be contacted to see if they retain any record of postoperative up to 30 day encounters and what the nature of the encounter was. Patients will NOT be contacted for the purpose of this QA study.

Approval for this study has been attained from the following:

1. University of British Columbia Research Ethics Board.
2. Vancouver Coastal Health Research Institute.

Study Personnel who will be retaining and invigilating patient charts will be the PI - a staff Anesthesiologist, a Resident in the UBC Anesthesiology Post-Graduate Program, and a UBC Medical Student.

It is anticipated that between 100 and 150 patients will have been through the STAR process at the time retrospective chart review begins.

ELIGIBILITY:
Inclusion Criteria:

* Surgical Team submits patient as potentially eligible for Same Day Discharge at the time of surgical booking.

Exclusion Criteria:

* Excluded if the patient never has a surgical procedure despite surgical booking and preoperative assessment. All patients must undergo surgery to be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hip joint pathology being booked for elective joint replacement by Orthopedics and earmarked by the surgeon as potentially Same Day Discharge eligible at the time of surgical booking.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
The number of patients who return to hospital for assessment and/or treatment of a surgical related problem or complication following Primary Total Hip Arthroplasty. | Within 30 days of elective Total Hip Arthroplasty surgery
  Patient records will be reviewed for hospital encounters within 30 days of their surgical procedure. If encounters are found within this timeframe, it will be discerned whether the encounter is for a surgically related problem or complication. Examples of surgically related problems include (but are not limited to) wound or surgical site infection, deep vein thrombosis, pulmonary embolism, pneumonia, urinary tract infection, pain issues as a result of having surgery, failure or concerns for the function of the new prosthesis, trauma or falls as a result of reduced mobility following surgery.

SECONDARY OUTCOMES:
The number of Patients who return to hospital for assessment and/or treatment of surgical related problems or complications following Primary Total Hip Arthroplasty. | Within 7 days of elective Total Hip Arthroplasty surgery
  Patient records will be reviewed for hospital encounters within 7 days of their surgical procedure. If encounters are found within this timeframe, it will be discerned whether the encounter is for a surgically related problem or complication in the same fashion as for the Primary Outcome Measure.

CONTACTS AND LOCATIONS:
Overall Officials: Donald J Young, MD, Principal Investigator — University of British Columbia, Vancouver Coastal Health
Locations (1):
- UBC Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meneghini R, Gibson W, Halsey D, Padgett D, Berend K, Della Valle CJ. The American Association of Hip and Knee Surgeons, Hip Society, Knee Society, and American Academy of Orthopaedic Surgeons Position Statement on Outpatient Joint Replacement. J Arthroplasty. 2018 Dec;33(12):3599-3601. doi: 10.1016/j.arth.2018.10.029. No abstract available. PMID 30449455
- [Background] Poitras S, Wood KS, Savard J, Dervin GF, Beaule PE. Predicting early clinical function after hip or knee arthroplasty. Bone Joint Res. 2015 Sep;4(9):145-51. doi: 10.1302/2046-3758.49.2000417. PMID 26336897
- [Background] Ziemba-Davis M, Caccavallo P, Meneghini RM. Outpatient Joint Arthroplasty-Patient Selection: Update on the Outpatient Arthroplasty Risk Assessment Score. J Arthroplasty. 2019 Jul;34(7S):S40-S43. doi: 10.1016/j.arth.2019.01.007. Epub 2019 Jan 15. PMID 30738619
- [Background] Meneghini RM, Ziemba-Davis M, Ishmael MK, Kuzma AL, Caccavallo P. Safe Selection of Outpatient Joint Arthroplasty Patients With Medical Risk Stratification: the "Outpatient Arthroplasty Risk Assessment Score". J Arthroplasty. 2017 Aug;32(8):2325-2331. doi: 10.1016/j.arth.2017.03.004. Epub 2017 Mar 14. PMID 28390881
- [Background] Sher A, Keswani A, Yao DH, Anderson M, Koenig K, Moucha CS. Predictors of Same-Day Discharge in Primary Total Joint Arthroplasty Patients and Risk Factors for Post-Discharge Complications. J Arthroplasty. 2017 Sep;32(9S):S150-S156.e1. doi: 10.1016/j.arth.2016.12.017. Epub 2016 Dec 22. PMID 28089186
- [Background] Kort NP, Bemelmans YFL, van der Kuy PHM, Jansen J, Schotanus MGM. Patient selection criteria for outpatient joint arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Sep;25(9):2668-2675. doi: 10.1007/s00167-016-4140-z. Epub 2016 Apr 22. PMID 27106923

DOCUMENTS (2):
  • Study Protocol (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT04120324/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT04120324/SAP_001.pdf